CLINICAL TRIAL: NCT02510573
Title: Prognostic Value of Serum Ficolin-3 Levels After Severe Traumatic Brain Injury：A Pilot Study
Brief Title: Low Serum Ficolin-3 Levels on Admission Are Associated With Poor Outcomes After Severe Traumatic Brain Injury
Status: Completed | Type: Observational
Sponsor: Sanmen People's Hospital (Other)
Responsible Party: Principal Investigator, Xiongwei Gao, Department of Neurosurgery, Sanmen People's Hospital
Other Study IDs: SM2015119
Record Dates: First submitted 2015-07-18; First posted 2015-07-29 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Brain Injuries
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — All blood samples from the patients at admission were collected in the tubes and centrifuged within 30 minutes at 1,000*g for 15 minutes. The serum was removed and frozen at -70°C until measurement.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- sTBI group: The patients with isolated head trauma and postresuscitation GCS score of 8 or less.

SUMMARY:
The current study was designed to investigate the change of serum ficolin-3 levels and assess the prognostic predictive effect of serum ficolin-3 levels in the patients with severe traumatic brain injury.

DETAILED DESCRIPTION:
Complement activation is one of the pathological mechanisms that contribute to the secondary brain injury after traumatic brain injury. Ficolin-mediated lectin pathways of complement activation contribute to the pathogenesis of ischemic stroke and may be additive to complement-independent inflammatory processes. Lower serum ficolin-3 levels have been demonstrated to be highly associated with unfavorable outcome after ischemic stroke. This prospective observatory study was designed to investigate the relationship between serum ficolin-3 levels and 1-week mortality, 6-month mortality and 6-month unfavorable outcome (defined as Glasgow Outcome Scale score of 1-3) in patients with severe traumatic brain injury. This study recruited 128 patients and 128 sex- and age- matched healthy controls. Serum ficolin-3 levels on admission were measured by sandwich immunoassays. It was postulated that serum ficolin-3 levels were correlated with Glasgow Coma Scale scores and ficolin-3 was identified as an independent prognostic predictor for 1-week mortality, 6-month mortality and 6-month unfavorable outcome. Thus, it was proposed that lower serum ficolin-3 levels, correlated with injury severity reflected by Glasgow Outcome Scale scores, had the potential to be the useful, complementary tool to predict short- or long- term clinical outcome after severe traumatic brain injury.

ELIGIBILITY:
Inclusion Criteria:

* Isolated head trauma
* Postresuscitation Glasgow Coma Scale score of 8 or less.

Exclusion Criteria:

* Less than 18 years of age
* Admission time > 6 hours
* Previous head trauma
* Neurological disease including ischemic or hemorrhagic stroke
* Use of antiplatelet or anticoagulant medication
* Diabetes mellitus
* Hypertension
* Presence of other prior systemic diseases including uremia, liver cirrhosis, malignancy, and chronic heart or lung disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients with isolated head trauma and postresuscitation Glasgow Coma Scale score of 8 or less.
Sampling Method: Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2011-04; Primary Completion 2014-07 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Mortality after severe traumatic brain injury | Follow-up of 6 months
  Using structure telephone interviews, follow-up was performed by 1 doctor who was blinded to clinical information.

SECONDARY OUTCOMES:
Unfavorable outcome after severe traumatic brain injury | Follow-up of 6 months
  Using structure telephone interviews, follow-up was performed by 1 doctor who was blinded to clinical information.